CLINICAL TRIAL: NCT00453986
Title: Lot-to-Lot Consistency, Non-Inferiority Versus Mencevax™ and Evaluation of the Co-Administration With Fluarix™ of GSK Biologicals' Meningococcal Vaccine GSK134612, in Healthy Subjects Aged 18 Through 55 Years of Age
Brief Title: Lot Consistency, Immuno, Safety of Meningococcal Vaccine GSK134612 Given With Fluarix™ to 18-55 Year-Old Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 109067
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Results first posted 2012-05-22 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2016-11

CONDITIONS: Infections, Meningococcal
Keywords: immunogenicity; Meningococcal serogroups A, C, W-135 and/or Y disease; co-administration; meningococcal vaccine; lot-to-lot consistency; conjugate vaccine
MeSH Terms: conditions — Meningococcal Infections | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- Nimenrix A Group (Experimental): subjects received 1 dose of Nimenrix™ Lot A at Month 0. Nimenrix™ vaccine was administered by intramuscular injection in the deltoid region of the non-dominant arm.
  Interventions: Biological: Meningococcal vaccine GSK134612
- Nimenrix B Group (Experimental): subjects received 1 dose of Nimenrix™ Lot B at Month 0. Nimenrix™ vaccine was administered by intramuscular injection in the deltoid region of the non-dominant arm.
  Interventions: Biological: Meningococcal vaccine GSK134612
- Nimenrix C Group (Experimental): subjects received 1 dose of Nimenrix™ Lot C at Month 0. Nimenrix™ vaccine was administered by intramuscular injection in the deltoid region of the non-dominant arm.
  Interventions: Biological: Meningococcal vaccine GSK134612
- Mencevax ACWY Group (Active Comparator): subjects received 1 dose of Mencevax™ ACWY vaccine at Month 0. Mencevax™ ACWY vaccine was administered by subcutaneous injection in the non-dominant upper arm.
  Interventions: Biological: Mencevax™ACWY
- Nimenrix+Fluarix Group (Experimental): subjects received 1 dose of Nimenrix™ Lot A co-administered with Fluarix™ vaccines at Month 0. Nimenrix™ vaccine was administered by intramuscular injection in the deltoid region of the non-dominant arm. Fluarix™ vaccine was administered by intramuscular injection in the deltoid region of the dominant arm.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Fluarix™

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — One intramuscular dose
  Arms: Nimenrix A Group; Nimenrix B Group; Nimenrix C Group; Nimenrix+Fluarix Group
Biological: Mencevax™ACWY — One subcutaneous dose
  Arms: Mencevax ACWY Group
Biological: Fluarix™ — One intramuscular dose
  Arms: Nimenrix+Fluarix Group

SUMMARY:
The purpose of this study is to demonstrate, in 18-55 year old adults, the consistency of different manufactured lots of meningococcal vaccine GSK134612, the non-inferiority of GSK134612 compared to licensed meningococcal vaccine Mencevax™, the non-inferiority of GSK134612 when given in an experimental co-administration with Fluarix™ compared to GSK134612 given alone and the immunogenicity of GSK134612 given with Fluarix™.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Multicentre study with 5 treatment groups. Three groups will receive three different manufactured lots of GSK134612, one group will receive one lot of GSK134612 given in an experimental co-administration with Fluarix™, the control group will receive Mencevax™. The study will be conducted in a double-blind manner with respect to the 3 lots of GSK134612 vaccine. The study will be 'open' between the groups receiving GSK134612 and the group receiving GSK134612 + Fluarix™ and the Mencevax™ group.

Each subject will have 2 blood samples taken for immunogenicity analyses, one prior to vaccination and one taken 30 days later.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 55 years of age at the time of the vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of his/her knowledge.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test, and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

For all subjects:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the dose of vaccine(s).
* Previous vaccination with meningococcal polysaccharide vaccine of serogroup A, C, W, and/or Y within the last five previous years.
* Previous vaccination with meningococcal polysaccharide conjugate vaccine of serogroup A, C, W, and/or Y.
* Previous vaccination with tetanus toxoid within the last month.
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Additional criteria for subjects receiving Fluarix™ co-administration:

* History of hypersensitivity to a previous dose of influenza vaccine.
* History of reactions or allergy likely to be exacerbated by any component of the vaccine including egg, chicken protein, formaldehyde, thimerosal, gentamicin sulfate, or sodium deoxycholate.
* History of administration of an influenza vaccine outside of this study, during current flu season.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1352 (Actual)
Dates: Start 2007-04-09; Primary Completion 2007-11-30 (Actual); Study Completion 2008-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Beirut, Lebanon
- Philippines (3):
  - GSK Investigational Site, Cavite
  - GSK Investigational Site, City of Muntinlupa
  - GSK Investigational Site, Manila

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dbaibo G, Macalalad N, Aplasca-De Los Reyes MR, Dimaano E, Bianco V, Baine Y, Miller J. The immunogenicity and safety of an investigational meningococcal serogroups A, C, W-135, Y tetanus toxoid conjugate vaccine (ACWY-TT) compared with a licensed meningococcal tetravalent polysaccharide vaccine: a randomized, controlled non-inferiority study. Hum Vaccin Immunother. 2012 Jul;8(7):873-80. doi: 10.4161/hv.20211. Epub 2012 Apr 9. PMID 22485050
- [Background] Macalalad N et al. The candidate Meningococcal serogroups A, C, W-135, Y conjugate vaccine (MenACWY-TT) and the seasonal influenza virus vaccine are immunogenic with an acceptable safety profile when co-administered in adults. Abstract presented at the 3rd Northern European Conference on Travel Medicine (NECTM) Hamburg, Germany, May 26-29, 2010.
- [Background] Aplasca-De Los Reyes MR, Dimaano E, Macalalad N, Dbaibo G, Bianco V, Baine Y, Miller J. The investigational meningococcal serogroups A, C, W-135, Y tetanus toxoid conjugate vaccine (ACWY-TT) and the seasonal influenza virus vaccine are immunogenic and well-tolerated when co-administered in adults. Hum Vaccin Immunother. 2012 Jul;8(7):881-7. doi: 10.4161/hv.20212. Epub 2012 Apr 9. PMID 22485048
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 109067 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109067 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109067 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109067 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109067 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109067 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109067 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were included in 1 of the 2 cohorts:
  Flu vaccine cohort: in the 5 groups, subjects received Nimenrix vaccine (lots A, B or C) or Mencevax ACWY vaccine or Nimenrix lot A and Fluarix vaccines.
  Non-Flu vaccine cohort: in the 4 groups, subjects received Nimenrix vaccine (lots A, B or C) or Mencevax ACWY vaccine.
Period: Overall Study
Arm/Group | Nimenrix A Group | Nimenrix B Group | Nimenrix C Group | Mencevax ACWY Group | Nimenrix+Fluarix Group
Started | 311 | 311 | 313 | 312 | 105
Completed | 305 | 306 | 307 | 310 | 105
Not Completed | 6 | 5 | 6 | 2 | 0
Not completed — Lost to Follow-up | 6 | 5 | 6 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix A Group | Nimenrix B Group | Nimenrix C Group | Mencevax ACWY Group | Nimenrix+Fluarix Group | Total
Number analyzed (Participants) | 311 | 311 | 313 | 312 | 105 | 1352
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.2 (10.48) | 35.1 (10.50) | 35.7 (10.75) | 34.9 (10.73) | 35.9 (10.40) | 35.4 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 139 | 133 | 151 | 40 | 598
  Male | 176 | 172 | 180 | 161 | 65 | 754
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South east Asian heritage | 223 | 223 | 224 | 224 | 105 | 999
  Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  White - Arabic / North African heritage | 88 | 88 | 87 | 88 | 0 | 351
  White - Caucasian / European heritage | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Serum Bactericidal Assay (Performed Using Baby Rabbit Complement) for Neisseria Meningitidis Serogroups A, C, W-135 and Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY) Antibody Titers, in Each of the 3 Lot Groups.
Description: Titers were expressed as geometric mean antibody titers and were calculated on all subjects from both cohorts receiving 1 dose of Nimenrix vaccine lot A, B or C.
Time Frame: One month after vaccination (at Month 1)
Population: The According-To-Protocol cohort for immunogenicity included all evaluable subjects from whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after the vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix A Group | Nimenrix B Group | Nimenrix C Group
Number analyzed (Participants) | 297 | 292 | 296
Titers
  rSBA-MenA: number analyzed (Participants) | 292 | 287 | 290
  rSBA-MenA | 3913.1 [3468.9 to 4414.1] | 3503.5 [3083.0 to 3981.4] | 3470.8 [3051.7 to 3947.3]
  rSBA-MenC: number analyzed (Participants) | 296 | 290 | 296
  rSBA-MenC | 9467.0 [7980.2 to 11230.7] | 8118.7 [6818.9 to 9666.3] | 9051.0 [7538.6 to 10866.8]
  rSBA-MenW-135 | 5263.2 [4527.0 to 6119.1] | 4890.6 [4145.5 to 5769.6] | 5260.1 [4536.8 to 6098.7]
  rSBA-MenY: number analyzed (Participants) | 297 | 292 | 295
  rSBA-MenY | 7872.7 [6849.0 to 9049.3] | 7235.7 [6257.6 to 8366.8] | 8041.4 [6952.1 to 9301.3]

2. Primary Outcome: Number of Subjects With a Vaccine Response for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Vaccine response was defined as a rSBA titer of at least 1:32 in initially seronegative subjects (<1:8) and as 4-fold increase in titer in initially seropositive subjects (≥1:8). A seronegative subject had antibody titer below 1:8 prior to vaccination and a seropositive subject had antibody titer equal to or above 1:8 prior to vaccination. Vaccine response was assessed for subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: One month after vaccination (at Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix Group: subjects received Nimenrix™ (Lots A without co-administration of Fluarix vaccine, B and C) at Month 0. Nimenrix™ vaccine was administered by intramuscular injection in the deltoid region of the non-dominant arm.
Arm/Group | Mencevax ACWY Group | Nimenrix Group
Number analyzed (Participants) | 288 | 862
Participants
  rSBA-MenA seronegative: number analyzed (Participants) | 25 | 109
  rSBA-MenA seronegative | 25 | 107
  rSBA-MenA seropositive: number analyzed (Participants) | 227 | 634
  rSBA-MenA seropositive | 151 | 488
  rSBA-MenC seronegative: number analyzed (Participants) | 66 | 200
  rSBA-MenC seronegative | 64 | 198
  rSBA-MenC seropositive: number analyzed (Participants) | 222 | 649
  rSBA-MenC seropositive | 201 | 579
  rSBA-MenW-135 seronegative: number analyzed (Participants) | 56 | 153
  rSBA-MenW-135 seronegative | 53 | 151
  rSBA-MenW-135 seropositive: number analyzed (Participants) | 227 | 707
  rSBA-MenW-135 seropositive | 189 | 625
  rSBA-MenY seronegative: number analyzed (Participants) | 32 | 70
  rSBA-MenY seronegative | 32 | 68
  rSBA-MenY seropositive: number analyzed (Participants) | 256 | 792
  rSBA-MenY seropositive | 195 | 682
  rSBA-MenA total: number analyzed (Participants) | 252 | 743
  rSBA-MenA total | 176 | 595
  rSBA-MenC total: number analyzed (Participants) | 288 | 849
  rSBA-MenC total | 265 | 777
  rSBA-MenW-135 total: number analyzed (Participants) | 283 | 860
  rSBA-MenW-135 total | 242 | 776
  rSBA-MenY total | 227 | 750

3. Primary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers, in Subjects Receiving the Nimenrix Lot A + Fluarix Vaccines or the Nimenrix Vaccine (Pooled Lots in the Flu Vaccine Cohort)
Description: Titers were expressed as geometric mean antibody titers and were calculated on all subjects receiving 1 dose of Nimenrix vaccine lot A co-administered with Fluarix vaccine and on subjects receiving 1 dose of Nimenrix vaccine among all the manufactured lots (pooled groups from the Flu vaccine cohort).
Time Frame: One month after vaccination (at Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Nimenrix (Flu Cohort) Group: Nimenrix A Group, Nimenrix B Group and Nimenrix C Group pooled groups from the Flu vaccine cohort. Nimenrix™ vaccine was administered by intramuscular injection in the deltoid region of the non-dominant arm.
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group
Number analyzed (Participants) | 105 | 308
Titers
  rSBA-MenA: number analyzed (Participants) | 102 | 306
  rSBA-MenA | 2831.1 [2282.4 to 3511.7] | 3784.2 [3326.3 to 4305.1]
  rSBA-MenC: number analyzed (Participants) | 105 | 306
  rSBA-MenC | 6579.5 [4861.5 to 8904.6] | 10130.8 [8672.3 to 11834.5]
  rSBA-MenW-135 | 4394.8 [3316.3 to 5824.0] | 6016.8 [5201.4 to 6960.2]
  rSBA-MenY: number analyzed (Participants) | 105 | 307
  rSBA-MenY | 5650.9 [4530.9 to 7047.] | 7464.1 [6500.3 to 8570.8]

4. Primary Outcome: Serum Haemagglutination Inhibition (HI) Antibody Titers Against Each of the 3 Influenza Virus Strains, in Subjects Receiving the Fluarix Vaccine.
Description: Titers were expressed as geometric mean antibody titers and were calculated on all subjects receiving 1 dose of Fluarix vaccine in the Flu vaccine cohort. The 3 influenza virus strains represented in the vaccine were A/H1N1, A/H3N2, and B.
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix+Fluarix Group
Number analyzed (Participants) | 105
Titers
  Anti-A/H1N1 [Month 0] | 54.1 [43.0 to 68.1]
  Anti-A/H1N1 [Month 1] | 537.2 [446.9 to 645.8]
  Anti-A/H3N2 [Month 0] | 31.5 [25.1 to 39.6]
  Anti-A/H3N2 [Month 1] | 177.8 [150.0 to 210.7]
  Anti-B [Month 0]: number analyzed (Participants) | 103
  Anti-B [Month 0] | 20.9 [17.0 to 25.7]
  Anti-B [Month 1]: number analyzed (Participants) | 104
  Anti-B [Month 1] | 192.7 [156.4 to 237.6]

5. Primary Outcome: Number of Seroconverted Subjects for HI Antibody Titers for Each of the 3 Influenza Virus Strains, in Subjects Receiving the Fluarix Vaccine.
Description: Seroconversion was defined as the percentage of subjects with either a pre-vaccination HI titer <1:10 and a post-vaccination titer >1:40, or a pre-vaccination titer >1:10 and a minimum 4-fold increase at post-vaccination titer, for each vaccine strain.
  Seroconversion was calculated on all subjects receiving 1 dose of Fluarix vaccine in the Flu vaccine cohort. The 3 influenza virus strains represented in the vaccine were A/H1N1, A/H3N2, and B.
Time Frame: One month after vaccination (at Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group
Number analyzed (Participants) | 105
Participants
  Anti-A/H1N1 | 75
  Anti-A/H3N2 | 65
  Anti-B: number analyzed (Participants) | 103
  Anti-B | 78

6. Primary Outcome: Seroconversion Factor for HI Antibody Titers for Each of the 3 Influenza Virus Strains, in Subjects Receiving the Fluarix Vaccine.
Description: Conversion factor defined as the fold increase in serum HI Geometric Mean Titers 1 month after vaccination compared to pre-vaccination, for each vaccine strain. Conversion factor was calculated on all subjects receiving 1 dose of Fluarix vaccine in the Flu vaccine cohort. The 3 influenza virus strains represented in the vaccine were A/H1N1, A/H3N2, and B.
Time Frame: One month after vaccination (at Month 1)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold increase in serum HI GMTs
Arm/Group | Nimenrix+Fluarix Group
Number analyzed (Participants) | 105
Fold increase in serum HI GMTs
  Anti-A/H1N1 | 9.9 [7.5 to 13.1]
  Anti-A/H3N2 | 5.6 [4.4 to 7.2]
  Anti-B: number analyzed (Participants) | 103
  Anti-B | 9.1 [7.1 to 11.6]

7. Primary Outcome: Number of Seroprotected Subjects HI Antibody Titers for Each of the 3 Influenza Virus Strains, in Subjects Receiving the Fluarix Vaccine.
Description: Seroprotection was defined as the percentage of subjects with a serum HI titer ≥ 1:40 after vaccination (for each vaccine strain) that usually is accepted as indicating protection. Seroprotection was calculated on all subjects receiving 1 dose of Fluarix vaccine in the Flu vaccine cohort. The 3 influenza virus strains represented in the vaccine were A/H1N1, A/H3N2, and B.
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group
Number analyzed (Participants) | 105
Participants
  Anti-A/H1N1 [Month 0] | 68
  Anti-A/H1N1 [Month 1] | 104
  Anti-A/H3N2 [Month 0] | 57
  Anti-A/H3N2 [Month 1] | 102
  Anti-B [Month 0]: number analyzed (Participants) | 103
  Anti-B [Month 0] | 44
  Anti-B [Month 1]: number analyzed (Participants) | 104
  Anti-B [Month 1] | 100

8. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135, and rSBA-MenY Titers Equal to or Above the Cut-off Values, in Each of the 3 Lot Groups.
Description: Assay cut-off values assessed were ≥1:8 and ≥1:128. Blood samples were taken on all subjects of both cohorts receiving 1 dose of Nimenrix vaccine lot A, B or C.
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix A Group | Nimenrix B Group | Nimenrix C Group
Number analyzed (Participants) | 297 | 292 | 296
Participants
  rSBA-MenA >= 1:8 [Month 0]: number analyzed (Participants) | 257 | 248 | 252
  rSBA-MenA >= 1:8 [Month 0] | 226 | 207 | 212
  rSBA-MenA >= 1:8 [Month 1]: number analyzed (Participants) | 292 | 287 | 290
  rSBA-MenA >= 1:8 [Month 1] | 292 | 287 | 289
  rSBA-MenC >= 1:8 [Month 0]: number analyzed (Participants) | 283 | 277 | 291
  rSBA-MenC >= 1:8 [Month 0] | 220 | 213 | 217
  rSBA-MenC >= 1:8 [Month 1]: number analyzed (Participants) | 296 | 290 | 296
  rSBA-MenC >= 1:8 [Month 1] | 296 | 289 | 295
  rSBA-MenW-135 >= 1:8 [Month 0]: number analyzed (Participants) | 287 | 286 | 287
  rSBA-MenW-135 >= 1:8 [Month 0] | 238 | 231 | 238
  rSBA-MenW-135 >= 1:8 [Month 1] | 297 | 290 | 296
  rSBA-MenY >= 1:8 [Month 0]: number analyzed (Participants) | 294 | 284 | 285
  rSBA-MenY >= 1:8 [Month 0] | 266 | 264 | 263
  rSBA-MenY >= 1:8 [Month 1]: number analyzed (Participants) | 297 | 292 | 295
  rSBA-MenY >= 1:8 [Month 1] | 297 | 291 | 294
  rSBA-MenA >= 1:128 [Month 0]: number analyzed (Participants) | 257 | 248 | 252
  rSBA-MenA >= 1:128 [Month 0] | 199 | 175 | 184
  rSBA-MenA >= 1:128 [Month 1]: number analyzed (Participants) | 292 | 287 | 290
  rSBA-MenA >= 1:128 [Month 1] | 291 | 286 | 288
  rSBA-MenC >= 1:128 [Month 0]: number analyzed (Participants) | 283 | 277 | 291
  rSBA-MenC >= 1:128 [Month 0] | 143 | 132 | 140
  rSBA-MenC >= 1:128 [Month 1]: number analyzed (Participants) | 296 | 290 | 296
  rSBA-MenC >= 1:128 [Month 1] | 293 | 286 | 293
  rSBA-MenW-135 >= 1:128 [Month 0]: number analyzed (Participants) | 287 | 286 | 287
  rSBA-MenW-135 >= 1:128 [Month 0] | 165 | 178 | 171
  rSBA-MenW-135 >= 1:128 [Month 1] | 294 | 289 | 295
  rSBA-MenY >= 1:128 [Month 0]: number analyzed (Participants) | 294 | 284 | 285
  rSBA-MenY >= 1:128 [Month 0] | 232 | 219 | 231
  rSBA-MenY >= 1:128 [Month 1]: number analyzed (Participants) | 297 | 292 | 295
  rSBA-MenY >= 1:128 [Month 1] | 295 | 291 | 293

9. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135, and rSBA-MenY Antibody Titers, in Each of the 3 Lot Groups.
Description: Titers were expressed as geometric mean antibody titers and were calculated on all subjects of both cohorts receiving 1 dose of Nimenrix vaccine lot A, B or C.
Time Frame: Prior to vaccination (at Month 0).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix A Group | Nimenrix B Group | Nimenrix C Group
Number analyzed (Participants) | 294 | 286 | 291
Titers
  rSBA-MenA [Month 0]: number analyzed (Participants) | 257 | 248 | 252
  rSBA-MenA [Month 0] | 215.1 [174.2 to 265.6] | 172.6 [135.9 to 219.2] | 157.5 [125.3 to 198.0]
  rSBA-MenC [Month 0]: number analyzed (Participants) | 283 | 277 | 291
  rSBA-MenC [Month 0] | 87.6 [69.2 to 110.9] | 83.2 [65.3 to 106.1] | 75.1 [59.5 to 94.7]
  rSBA-MenW-135 [Month 0]: number analyzed (Participants) | 287 | 286 | 287
  rSBA-MenW-135 [Month 0] | 111.7 [90.3 to 138.2] | 124.6 [98.8 to 157.2] | 115.1 [92.4 to 143.5]
  rSBA-MenY [Month 0]: number analyzed (Participants) | 294 | 284 | 285
  rSBA-MenY [Month 0] | 275.8 [224.8 to 338.4] | 270.3 [223.6 to 326.7] | 315.6 [260.6 to 382.1]

10. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135, and rSBA-MenY Titers Equal to or Above the Cut-off Values, for Subjects in the Flu Vaccine Cohort
Description: Assay cut-off values assessed were ≥1:8 and ≥1:128. Blood samples were taken on all subjects receiving 1 dose of Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving 1 dose of Nimenrix vaccine among all the manufactured lots (pooled groups from the Flu vaccine cohort) and on subjects receiving 1 dose of Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Mencevax ACWY (Flu Cohort) Group: Mencevax ACWY Group from the Flu vaccine cohort. MencevaxTM ACWY vaccine was administered by subcutaneous injection in the non-dominant upper arm.
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 308 | 104
Participants
  rSBA-MenA >=1:8 [Month 0]: number analyzed (Participants) | 88 | 265 | 88
  rSBA-MenA >=1:8 [Month 0] | 81 | 219 | 82
  rSBA-MenA >=1:8 [Month 1]: number analyzed (Participants) | 102 | 306 | 104
  rSBA-MenA >=1:8 [Month 1] | 102 | 305 | 104
  rSBA-MenC >=1:8 [Month 0]: number analyzed (Participants) | 97 | 294 | 101
  rSBA-MenC >=1:8 [Month 0] | 84 | 225 | 84
  rSBA-MenC >=1:8 [Month 1]: number analyzed (Participants) | 105 | 306 | 104
  rSBA-MenC >=1:8 [Month 1] | 104 | 306 | 103
  rSBA-MenW-135 >=1:8 [Month 0]: number analyzed (Participants) | 101 | 299 | 102
  rSBA-MenW-135 >=1:8 [Month 0] | 85 | 259 | 84
  rSBA-MenW-135 >=1:8 [Month 1] | 105 | 308 | 103
  rSBA-MenY >=1:8 [Month 0]: number analyzed (Participants) | 102 | 301 | 100
  rSBA-MenY >=1:8 [Month 0] | 96 | 277 | 88
  rSBA-MenY >=1:8 [Month 1]: number analyzed (Participants) | 105 | 307 | 104
  rSBA-MenY >=1:8 [Month 1] | 105 | 306 | 104
  rSBA-MenA >=1:128 [Month 0]: number analyzed (Participants) | 88 | 265 | 88
  rSBA-MenA >=1:128 [Month 0] | 64 | 180 | 69
  rSBA-MenA >=1:128 [Month 1]: number analyzed (Participants) | 102 | 306 | 104
  rSBA-MenA >=1:128 [Month 1] | 101 | 305 | 103
  rSBA-MenC >=1:128 [Month 0]: number analyzed (Participants) | 97 | 294 | 101
  rSBA-MenC >=1:128 [Month 0] | 58 | 154 | 54
  rSBA-MenC >=1:128 [Month 1]: number analyzed (Participants) | 105 | 306 | 104
  rSBA-MenC >=1:128 [Month 1] | 103 | 304 | 103
  rSBA-MenW-135 >=1:128 [Month 0]: number analyzed (Participants) | 101 | 299 | 102
  rSBA-MenW-135 >=1:128 [Month 0] | 62 | 192 | 54
  rSBA-MenW-135 >=1:128 [Month 1] | 102 | 306 | 102
  rSBA-MenY >=1:128 [Month 0]: number analyzed (Participants) | 102 | 301 | 100
  rSBA-MenY >=1:128 [Month 0] | 82 | 228 | 79
  rSBA-MenY >=1:128 [Month 1]: number analyzed (Participants) | 105 | 307 | 104
  rSBA-MenY >=1:128 [Month 1] | 104 | 305 | 103

11. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135, and rSBA-MenY Antibody Titers, for Subjects in the Flu Vaccine Cohort
Description: Titers were expressed as geometric mean antibody titers and were calculated on all subjects receiving 1 dose of Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving 1 dose of Nimenrix vaccine among all the manufactured lots (pooled groups from the Flu vaccine cohort) and on subjects receiving 1 dose of Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 308 | 104
Titers
  rSBA-MenA [Month 0]: number analyzed (Participants) | 88 | 265 | 88
  rSBA-MenA [Month 0] | 200.5 [145.3 to 276.8] | 154.8 [122.2 to 196.1] | 250.8 [182.0 to 345.6]
  rSBA-MenA [Month 1]: number analyzed (Participants) | 102 | 306 | 104
  rSBA-MenA [Month 1] | 2831.1 [2282.4 to 3511.7] | 3784.2 [3326.3 to 4305.1] | 1826.9 [1492.3 to 2236.6]
  rSBA-MenC [Month 0]: number analyzed (Participants) | 97 | 294 | 101
  rSBA-MenC [Month 0] | 139.1 [94.2 to 205.2] | 100.8 [78.4 to 129.6] | 120.0 [78.7 to 182.8]
  rSBA-MenC [Month 1]: number analyzed (Participants) | 105 | 306 | 104
  rSBA-MenC [Month 1] | 6579.5 [4861.5 to 8904.6] | 10130.8 [8672.3 to 11834.5] | 8784.9 [6759.4 to 11417.3]
  rSBA-MenW-135 [Month 0]: number analyzed (Participants) | 101 | 299 | 102
  rSBA-MenW-135 [Month 0] | 121.0 [84.3 to 173.7] | 146.2 [119.5 to 178.8] | 86.2 [60.9 to 121.9]
  rSBA-MenW-135 [Month 1] | 4394.8 [3316.3 to 5824.0] | 6016.8 [5201.4 to 6960.2] | 2361.1 [1757.7 to 3171.6]
  rSBA-MenY [Month 0]: number analyzed (Participants) | 102 | 301 | 100
  rSBA-MenY [Month 0] | 309.6 [229.9 to 417.0] | 287.4 [236.2 to 349.6] | 209.9 [147.4 to 299.0]
  rSBA-MenY [Month 1]: number analyzed (Participants) | 105 | 307 | 104
  rSBA-MenY [Month 1] | 5650.9 [4530.9 to 7047.7] | 7464.1 [6500.3 to 8570.8] | 3363.5 [2630.9 to 4300.1]

12. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135, and rSBA-MenY Titers Equal to or Above the Cut-off Values, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Assay cut-off values assessed were ≥1:8 and ≥1:128. Blood samples were taken on all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix Group: subjects received Nimenrix™ (Lots A without co-administration of FluarixTM vaccine, B and C) at Month 0. Nimenrix™ vaccine was administered by intramuscular injection in the deltoid region of the non-dominant arm.
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 885 | 294
Participants
  rSBA-MenA >=1:8 [Month 0]: number analyzed (Participants) | 757 | 254
  rSBA-MenA >=1:8 [Month 0] | 645 | 229
  rSBA-MenA >=1:8 [Month 1]: number analyzed (Participants) | 869 | 291
  rSBA-MenA >=1:8 [Month 1] | 868 | 291
  rSBA-MenC >=1:8 [Month 0]: number analyzed (Participants) | 851 | 289
  rSBA-MenC >=1:8 [Month 0] | 650 | 223
  rSBA-MenC >=1:8 [Month 1]: number analyzed (Participants) | 882 | 293
  rSBA-MenC >=1:8 [Month 1] | 880 | 291
  rSBA-MenW-135 >=1:8 [Month 0]: number analyzed (Participants) | 860 | 283
  rSBA-MenW-135 >=1:8 [Month 0] | 707 | 227
  rSBA-MenW-135 >=1:8 [Month 1] | 883 | 292
  rSBA-MenY >=1:8 [Month 0]: number analyzed (Participants) | 863 | 288
  rSBA-MenY >=1:8 [Month 0] | 793 | 256
  rSBA-MenY >=1:8 [Month 1]: number analyzed (Participants) | 884 | 294
  rSBA-MenY >=1:8 [Month 1] | 882 | 294
  rSBA-MenA >=1:128 [Month 0]: number analyzed (Participants) | 757 | 254
  rSBA-MenA >=1:128 [Month 0] | 558 | 200
  rSBA-MenA >=1:128 [Month 1]: number analyzed (Participants) | 869 | 291
  rSBA-MenA >=1:128 [Month 1] | 865 | 290
  rSBA-MenC >=1:128 [Month 0]: number analyzed (Participants) | 851 | 289
  rSBA-MenC >=1:128 [Month 0] | 415 | 152
  rSBA-MenC >=1:128 [Month 1]: number analyzed (Participants) | 882 | 293
  rSBA-MenC >=1:128 [Month 1] | 872 | 289
  rSBA-MenW-135 >=1:128 [Month 0]: number analyzed (Participants) | 860 | 283
  rSBA-MenW-135 >=1:128 [Month 0] | 514 | 155
  rSBA-MenW-135 >=1:128 [Month 1] | 878 | 288
  rSBA-MenY >=1:128 [Month 0]: number analyzed (Participants) | 863 | 288
  rSBA-MenY >=1:128 [Month 0] | 682 | 224
  rSBA-MenY >=1:128 [Month 1]: number analyzed (Participants) | 884 | 294
  rSBA-MenY >=1:128 [Month 1] | 879 | 293

13. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135, and rSBA-MenY Antibody Titers, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Titers were expressed as geometric mean antibody titers and were calculated on all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 885 | 294
Titers
  rSBA-MenA [Month 0]: number analyzed (Participants) | 757 | 254
  rSBA-MenA [Month 0] | 180.4 [158.4 to 205.6] | 216.3 [177.4 to 263.7]
  rSBA-MenA [Month 1]: number analyzed (Participants) | 869 | 291
  rSBA-MenA [Month 1] | 3624.7 [3371.7 to 3896.8] | 2127.2 [1909.2 to 2370.1]
  rSBA-MenC [Month 0]: number analyzed (Participants) | 851 | 289
  rSBA-MenC [Month 0] | 81.7 [71.3 to 93.7] | 91.2 [71.5 to 116.4]
  rSBA-MenC [Month 1]: number analyzed (Participants) | 882 | 293
  rSBA-MenC [Month 1] | 8865.9 [8011.0 to 9812.0] | 7371.2 [6297.4 to 8628.2]
  rSBA-MenW-135 [Month 0]: number analyzed (Participants) | 860 | 283
  rSBA-MenW-135 [Month 0] | 117.0 [103.0 to 132.9] | 94.0 [75.2 to 117.4]
  rSBA-MenW-135 [Month 1] | 5136.2 [4698.8 to 5614.3] | 2461.3 [2081.0 to 2911.0]
  rSBA-MenY [Month 0]: number analyzed (Participants) | 863 | 288
  rSBA-MenY [Month 0] | 286.5 [256.0 to 320.6] | 262.2 [211.8 to 324.5]
  rSBA-MenY [Month 1]: number analyzed (Participants) | 884 | 294
  rSBA-MenY [Month 1] | 7710.7 [7100.1 to 8373.8] | 4314.3 [3782.1 to 4921.5]

14. Secondary Outcome: Number of Subjects With a Vaccine Response for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody, for Subjects in the Flu Vaccine Cohort
Description: Vaccine response was defined as a rSBA titer of at least 1:32 in initially seronegative subjects (<1:8) and as 4-fold increase in titer in initially seropositive subjects (≥ 1:8). A seronegative subject had antibody titer >1:8 and a seropositive subject had antibody titer ≥1:8 prior to vaccination. Vaccine response was assessed for subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: One month after vaccination (at Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 102 | 300 | 102
Participants
  rSBA-MenA seronegative: number analyzed (Participants) | 5 | 45 | 6
  rSBA-MenA seronegative | 5 | 44 | 6
  rSBA-MenA seropositive: number analyzed (Participants) | 80 | 218 | 82
  rSBA-MenA seropositive | 60 | 168 | 50
  rSBA-MenC seronegative: number analyzed (Participants) | 13 | 68 | 17
  rSBA-MenC seronegative | 13 | 68 | 16
  rSBA-MenC seropositive: number analyzed (Participants) | 84 | 225 | 84
  rSBA-MenC seropositive | 73 | 193 | 72
  rSBA-MenW-135 seronegative: number analyzed (Participants) | 16 | 40 | 18
  rSBA-MenW-135 seronegative | 15 | 40 | 17
  rSBA-MenW-135 seropositive: number analyzed (Participants) | 85 | 259 | 84
  rSBA-MenW-135 seropositive | 74 | 235 | 72
  rSBA-MenY seronegative: number analyzed (Participants) | 6 | 24 | 12
  rSBA-MenY seronegative | 6 | 23 | 12
  rSBA-MenY seropositive: number analyzed (Participants) | 96 | 276 | 88
  rSBA-MenY seropositive | 77 | 236 | 61
  rSBA-MenA total: number analyzed (Participants) | 85 | 263 | 88
  rSBA-MenA total | 65 | 212 | 56
  rSBA-MenC total: number analyzed (Participants) | 97 | 293 | 101
  rSBA-MenC total | 86 | 261 | 88
  rSBA-MenW-135 total: number analyzed (Participants) | 101 | 299 | 102
  rSBA-MenW-135 total | 89 | 275 | 89
  rSBA-MenY total: number analyzed (Participants) | 102 | 300 | 100
  rSBA-MenY total | 83 | 259 | 73

15. Secondary Outcome: Number of Subjects With Anti-tetanus Antibody Concentrations Equal to or Above the Cut-off Value of 0.1 International Unit Per Milliliter (IU/mL), in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Blood samples were taken on all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 885 | 293
Participants
  Anti-tetanus [Month 0]: number analyzed (Participants) | 882 | 293
  Anti-tetanus [Month 0] | 454 | 153
  Anti-tetanus [Month 1] | 703 | 156

16. Secondary Outcome: Anti-tetanus Antibody Concentrations, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Concentrations were expressed in geometric mean concentrations in International unit per milliliter (IU/mL) and were calculated on all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 885 | 293
IU/mL
  Anti-tetanus [Month 0]: number analyzed (Participants) | 882 | 293
  Anti-tetanus [Month 0] | 0.245 [0.217 to 0.277] | 0.265 [0.214 to 0.329]
  Anti-tetanus [Month 1] | 3.488 [2.949 to 4.126] | 0.279 [0.224 to 0.347]

17. Secondary Outcome: Number of Subjects With Anti-tetanus Antibody Concentrations Equal to or Above the Cut-off Value of 0.1 International Unit Per Milliliter (IU/mL), for Subjects in the Flu Vaccine Cohort
Description: Blood samples were taken on subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 308 | 104
Participants
  Anti-tetanus [Month 0]: number analyzed (Participants) | 105 | 308 | 103
  Anti-tetanus [Month 0] | 61 | 193 | 54
  Anti-tetanus [Month 1] | 84 | 254 | 53

18. Secondary Outcome: Anti-tetanus Antibody Concentrations for Subjects in the Flu Vaccine Cohort
Description: Concentrations were expressed in geometric mean concentrations in International unit per milliliter (IU/mL) and were calculated on subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 308 | 104
IU/mL
  Anti-tetanus [Month 0]: number analyzed (Participants) | 105 | 308 | 103
  Anti-tetanus [Month 0] | 0.295 [0.206 to 0.421] | 0.418 [0.334 to 0.523] | 0.287 [0.197 to 0.419]
  Anti-tetanus [Month 1] | 3.073 [1.937 to 4.874] | 4.655 [3.557 to 6.092] | 0.276 [0.190 to 0.402]

19. Secondary Outcome: Number of Subjects With Anti-meningococcal Polysaccharide Serogroups, A, C, W-135 and Y Antibody Concentrations Equal to or Above the Cut-off Values, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Meningococcal polysaccharide serogroups, A, C, W-135 and Y = PSA, PSC, PSW-135 & PSY. Assay cut-off values assessed were ≥ 0.3 microgram per milliliter (µg/mL) and ≥ 2.0 µg/mL. Blood samples were taken on all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 449 | 148
Participants
  Anti-PSA >=0.3 µg/mL [Month 0]: number analyzed (Participants) | 413 | 141
  Anti-PSA >=0.3 µg/mL [Month 0] | 354 | 125
  Anti-PSA >=0.3 µg/mL [Month 1]: number analyzed (Participants) | 432 | 144
  Anti-PSA >=0.3 µg/mL [Month 1] | 432 | 144
  Anti-PSC >=0.3 µg/mL [Month 0]: number analyzed (Participants) | 427 | 139
  Anti-PSC >=0.3 µg/mL [Month 0] | 130 | 61
  Anti-PSC >=0.3 µg/mL [Month 1]: number analyzed (Participants) | 425 | 142
  Anti-PSC >=0.3 µg/mL [Month 1] | 422 | 141
  Anti-PSW-135 >=0.3 µg/mL [Month 0]: number analyzed (Participants) | 416 | 144
  Anti-PSW-135 >=0.3 µg/mL [Month 0] | 135 | 38
  Anti-PSW-135 >=0.3 µg/mL [Month 1]: number analyzed (Participants) | 449 | 146
  Anti-PSW-135 >=0.3 µg/mL [Month 1] | 439 | 144
  Anti-PSY >=0.3 µg/mL [Month 0]: number analyzed (Participants) | 424 | 143
  Anti-PSY >=0.3 µg/mL [Month 0] | 156 | 52
  Anti-PSY >=0.3 µg/mL [Month 1] | 442 | 145
  Anti-PSA >=2.0 µg/mL [Month 0]: number analyzed (Participants) | 413 | 141
  Anti-PSA >=2.0 µg/mL [Month 0] | 227 | 87
  Anti-PSA >=2.0 µg/mL [Month 1]: number analyzed (Participants) | 432 | 144
  Anti-PSA >=2.0 µg/mL [Month 1] | 428 | 144
  Anti-PSC >=2.0 µg/mL [Month 0]: number analyzed (Participants) | 427 | 139
  Anti-PSC >=2.0 µg/mL [Month 0] | 51 | 17
  Anti-PSC >=2.0 µg/mL [Month 1]: number analyzed (Participants) | 425 | 142
  Anti-PSC >=2.0 µg/mL [Month 1] | 398 | 141
  Anti-PSW-135 >=2.0 µg/mL [Month 0]: number analyzed (Participants) | 416 | 144
  Anti-PSW-135 >=2.0 µg/mL [Month 0] | 41 | 11
  Anti-PSW-135 >=2.0 µg/mL [Month 1]: number analyzed (Participants) | 449 | 146
  Anti-PSW-135 >=2.0 µg/mL [Month 1] | 408 | 136
  Anti-PSY >=2.0 µg/mL [Month 0]: number analyzed (Participants) | 424 | 143
  Anti-PSY >=2.0 µg/mL [Month 0] | 59 | 21
  Anti-PSY >=2.0 µg/mL [Month 1] | 420 | 142

20. Secondary Outcome: Anti-PSA, Anti-PSC, Anti-PSW-135 & Anti-PSY Antibody Concentrations, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Concentrations were expressed in geometric mean concentrations in microgram per milliliter (µg/mL) and were calculated on all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 449 | 148
µg/mL
  Anti-PSA [Month 0]: number analyzed (Participants) | 413 | 141
  Anti-PSA [Month 0] | 2.14 [1.82 to 2.52] | 2.65 [2.05 to 3.43]
  Anti-PSA [Month 1]: number analyzed (Participants) | 432 | 144
  Anti-PSA [Month 1] | 101.79 [88.95 to 116.49] | 56.89 [46.73 to 69.26]
  Anti-PSC [Month 0]: number analyzed (Participants) | 427 | 139
  Anti-PSC [Month 0] | 0.33 [0.29 to 0.37] | 0.38 [0.30 to 0.49]
  Anti-PSC [Month 1]: number analyzed (Participants) | 425 | 142
  Anti-PSC [Month 1] | 20.96 [18.26 to 24.05] | 45.85 [37.97 to 55.35]
  Anti-PSW-135 [Month 0]: number analyzed (Participants) | 416 | 144
  Anti-PSW-135 [Month 0] | 0.31 [0.27 to 0.35] | 0.26 [0.22 to 0.30]
  Anti-PSW-135 [Month 1]: number analyzed (Participants) | 449 | 146
  Anti-PSW-135 [Month 1] | 24.71 [20.75 to 29.42] | 21.90 [16.86 to 28.44]
  Anti-PSY [Month 0]: number analyzed (Participants) | 424 | 143
  Anti-PSY [Month 0] | 0.36 [0.32 to 0.41] | 0.35 [0.28 to 0.44]
  Anti-PSY [Month 1] | 36.94 [31.10 to 43.87] | 30.41 [22.94 to 40.30]

21. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW-135 & Anti-PSY Antibody Concentrations Equal to or Above the Cut-off Values, for Subjects in the Flu Vaccine Cohort
Description: Assay cut-off values assessed were ≥ 0.3 microgram per milliliter (µg/mL) and ≥ 2.0 µg/mL. Blood samples were taken on subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 54 | 157 | 52
Participants
  Anti-PSA >=0.3 µg/mL [Month 0]: number analyzed (Participants) | 50 | 143 | 52
  Anti-PSA >=0.3 µg/mL [Month 0] | 46 | 136 | 51
  Anti-PSA >=0.3 µg/mL [Month 1]: number analyzed (Participants) | 50 | 151 | 52
  Anti-PSA >=0.3 µg/mL [Month 1] | 49 | 151 | 52
  Anti-PSC >=0.3 µg/mL [Month 0]: number analyzed (Participants) | 51 | 149 | 50
  Anti-PSC >=0.3 µg/mL [Month 0] | 16 | 50 | 24
  Anti-PSC >=0.3 µg/mL [Month 1]: number analyzed (Participants) | 49 | 146 | 52
  Anti-PSC >=0.3 µg/mL [Month 1] | 48 | 145 | 51
  Anti-PSW-135 >=0.3 µg/mL [Month 0]: number analyzed (Participants) | 47 | 144 | 48
  Anti-PSW-135 >=0.3 µg/mL [Month 0] | 12 | 53 | 11
  Anti-PSW-135 >=0.3 µg/mL [Month 1]: number analyzed (Participants) | 53 | 157 | 49
  Anti-PSW-135 >=0.3 µg/mL [Month 1] | 51 | 153 | 49
  Anti-PSY >=0.3 µg/mL [Month 0]: number analyzed (Participants) | 51 | 147 | 50
  Anti-PSY >=0.3 µg/mL [Month 0] | 13 | 61 | 17
  Anti-PSY >=0.3 µg/mL [Month 1] | 53 | 156 | 51
  Anti-PSA >=2.0 µg/mL [Month 0]: number analyzed (Participants) | 50 | 143 | 52
  Anti-PSA >=2.0 µg/mL [Month 0] | 30 | 100 | 37
  Anti-PSA >=2.0 µg/mL [Month 1]: number analyzed (Participants) | 50 | 151 | 52
  Anti-PSA >=2.0 µg/mL [Month 1] | 49 | 149 | 52
  Anti-PSC >=2.0 µg/mL [Month 0]: number analyzed (Participants) | 51 | 149 | 50
  Anti-PSC >=2.0 µg/mL [Month 0] | 5 | 24 | 8
  Anti-PSC >=2.0 µg/mL [Month 1]: number analyzed (Participants) | 49 | 146 | 52
  Anti-PSC >=2.0 µg/mL [Month 1] | 42 | 133 | 51
  Anti-PSW-135 >=2.0 µg/mL [Month 0]: number analyzed (Participants) | 47 | 144 | 48
  Anti-PSW-135 >=2.0 µg/mL [Month 0] | 1 | 13 | 4
  Anti-PSW-135 >=2.0 µg/mL [Month 1]: number analyzed (Participants) | 53 | 157 | 49
  Anti-PSW-135 >=2.0 µg/mL [Month 1] | 46 | 142 | 48
  Anti-PSY >=2.0 µg/mL [Month 0]: number analyzed (Participants) | 51 | 147 | 50
  Anti-PSY >=2.0 µg/mL [Month 0] | 6 | 25 | 6
  Anti-PSY >=2.0 µg/mL [Month 1] | 51 | 147 | 50

22. Secondary Outcome: Anti-PSA, Anti-PSC, Anti-PSW-135 & Anti-PSY Antibody Concentrations, for Subjects in the Flu Vaccine Cohort
Description: Concentrations were expressed in geometric mean concentrations in microgram per milliliter (µg/mL) and were calculated on subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: Prior to and one month after vaccination (at Month 0 and Month 1).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 54 | 157 | 52
µg/mL
  Anti-PSA [Month 0]: number analyzed (Participants) | 50 | 143 | 52
  Anti-PSA [Month 0] | 2.40 [1.61 to 3.58] | 4.08 [3.16 to 5.26] | 3.83 [2.64 to 5.56]
  Anti-PSA [Month 1]: number analyzed (Participants) | 50 | 151 | 52
  Anti-PSA [Month 1] | 56.47 [35.76 to 89.19] | 142.33 [113.63 to 178.28] | 56.43 [40.72 to 78.18]
  Anti-PSC [Month 0]: number analyzed (Participants) | 51 | 149 | 50
  Anti-PSC [Month 0] | 0.30 [0.22 to 0.41] | 0.41 [0.31 to 0.53] | 0.48 [0.30 to 0.76]
  Anti-PSC [Month 1]: number analyzed (Participants) | 49 | 146 | 52
  Anti-PSC [Month 1] | 9.05 [5.70 to 14.36] | 19.26 [15.22 to 24.37] | 46.30 [32.29 to 66.39]
  Anti-PSW-135 [Month 0]: number analyzed (Participants) | 47 | 144 | 48
  Anti-PSW-135 [Month 0] | 0.21 [0.18 to 0.26] | 0.33 [0.27 to 0.40] | 0.25 [0.18 to 0.35]
  Anti-PSW-135 [Month 1]: number analyzed (Participants) | 53 | 157 | 49
  Anti-PSW-135 [Month 1] | 20.06 [12.27 to 32.81] | 26.44 [19.66 to 35.55] | 26.27 [17.54 to 39.35]
  Anti-PSY [Month 0]: number analyzed (Participants) | 51 | 147 | 50
  Anti-PSY [Month 0] | 0.29 [0.20 to 0.43] | 0.41 [0.32 to 0.52] | 0.32 [0.22 to 0.46]
  Anti-PSY [Month 1] | 25.39 [15.71 to 41.01] | 40.46 [30.00 to 54.57] | 24.67 [15.03 to 40.51]

23. Secondary Outcome: Number of Subjects With Any and Severe Solicited Local Symptoms, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any solicited local symptom irrespective of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling above 50 millimeter (mm). Solicited local symptoms were collected for all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: During the 4-day (Days 0-3) follow-up period after vaccination
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 927 | 310
Participants
  Any pain | 180 | 42
  Grade 3 pain | 4 | 1
  Any redness | 82 | 14
  Redness > 50 mm | 12 | 0
  Any swelling | 73 | 6
  Swelling > 50 mm | 10 | 0

24. Secondary Outcome: Number of Subjects With Any and Severe Solicited Local Symptoms, for Subjects in the Flu Vaccine Cohort Receiving the Nimenrix or the Mencevax ACWY Vaccines.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any solicited local symptom irrespective of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling above 50 millimeter (mm). Solicited local symptoms were collected for subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: During the 4-day (Days 0-3) follow-up period after meningococcal vaccination
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 311 | 104
Participants
  Any pain | 23 | 84 | 16
  Grade 3 pain | 1 | 0 | 0
  Any redness | 6 | 38 | 5
  Redness > 50 mm | 0 | 1 | 0
  Any swelling | 4 | 32 | 1
  Swelling > 50 mm | 0 | 3 | 0

25. Secondary Outcome: Number of Subjects With Any and Severe Solicited Local Symptoms, in Subjects Receiving the Fluarix Vaccine
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any solicited local symptom irrespective of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling above 50 millimeter (mm). Solicited local symptoms were collected for subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine after the Fluarix vaccine administration.
Time Frame: During the 4-day (Days 0-3) follow-up period after Fluarix vaccine administration
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group
Number analyzed (Participants) | 105
Participants
  Any pain | 29
  Grade 3 pain | 1
  Any redness | 7
  Redness > 50 mm | 0
  Any swelling | 7
  Swelling > 50 mm | 1

26. Secondary Outcome: Number of Subjects With Any and Severe Solicited General Symptoms, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache and fever (= axillary temperature ≥ 37.5 degrees Celsius). Any = occurrence of any solicited general symptom irrespective of intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal activities. Grade 3 fever = axillary temperature > 39.5°C. Symptoms were collected for all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: During the 4-day (Days 0-3) follow-up period after vaccination
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 927 | 310
Participants
  Any fatigue | 114 | 30
  Grade 3 fatigue | 8 | 0
  Fever >= 37.5°C | 37 | 14
  Fever > 39.5°C | 2 | 2
  Any gastrointestinal symptoms | 43 | 10
  Grade 3 gastrointestinal symptoms | 2 | 1
  Any headache | 151 | 44
  Grade 3 headache | 14 | 5

27. Secondary Outcome: Number of Subjects With Any and Severe Solicited General Symptoms, for Subjects in the Flu Vaccine Cohort
Description: Solicited general symptoms = fatigue, gastrointestinal symptoms, headache and fever (= axillary temperature ≥ 37.5°C). Any = occurrence of any solicited general symptom irrespective of intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal activities. Grade 3 fever = > 39.5°C. Symptoms were collected for subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: During the 4-day (Days 0-3) follow-up period after vaccination
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 311 | 104
Participants
  Any fatigue | 10 | 33 | 12
  Grade 3 fatigue | 0 | 0 | 0
  Fever >= 37.5°C | 3 | 10 | 3
  Fever > 39.5°C | 0 | 1 | 0
  Any gastrointestinal symptoms | 2 | 15 | 2
  Grade 3 gastrointestinal symptoms | 0 | 0 | 0
  Any headache | 14 | 47 | 12
  Grade 3 headache | 0 | 1 | 0

28. Secondary Outcome: Number of Subjects Reporting Rash, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: Rash assessed were hives, idiopathic thrombocytopenic purpura and petechiae and were collected for all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: From Dose 1 (at Month 0) up to study end (at Month 6)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 935 | 312
Participants | 10 | 3

29. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Illness(es) (NOCIs), in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: NOCIs assessed were autoimmune disorders, asthma, type I diabetes and allergies and were collected for all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: From Dose 1 (at Month 0) up to study end (at Month 6)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 935 | 312
Participants | 0 | 0

30. Secondary Outcome: Number of Subjects Reporting Adverse Events (AEs) Resulting in Emergency Room (ER) Visits, in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: AEs resulting in ER visits were collected for all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: From Dose 1 (at Month 0) up to study end (at Month 6)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 935 | 312
Participants | 13 | 1

31. Secondary Outcome: Number of Subjects Reporting Rash, for Subjects in the Flu Vaccine Cohort
Description: Rash assessed were hives, idiopathic thrombocytopenic purpura and petechiae and were collected for subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: From Dose 1 (at Month 0) up to study end (at Month 6)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 311 | 104
Participants | 0 | 3 | 0

32. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Illness(es) (NOCIs), for Subjects in the Flu Vaccine Cohort
Description: NOCIs assessed were autoimmune disorders, asthma, type I diabetes and allergies and were collected for subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: From Dose 1 (at Month 0) up to study end (at Month 6)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 311 | 104
Participants | 0 | 0 | 0

33. Secondary Outcome: Number of Subjects Reporting Adverse Events (AEs) Resulting in Emergency Room (ER) Visits, for Subjects in the Flu Vaccine Cohort
Description: AEs resulting in ER visits were collected for subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: From Dose 1 (at Month 0) up to study end (at Month 6)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 311 | 104
Participants | 0 | 0 | 0

34. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs), in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Unsolicited AEs were collected for all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, B and C) or the Mencevax ACWY vaccine.
Time Frame: From Dose 1 (at Month 0) up to 1 month after vaccination (at Month 1)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 935 | 312
Participants | 135 | 47

35. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs), in Subjects Receiving the Nimenrix (From the 3 Manufactured Lots Pooled) or the Mencevax ACWY Vaccines.
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. SAEs were collected for all subjects of both cohorts receiving the Nimenrix vaccine (lot A without co-administration of Fluarix vaccine, lot B and lot C) or the Mencevax ACWY vaccine.
Time Frame: From Dose 1 (at Month 0) up to study end (at Month 6)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 935 | 312
Participants | 7 | 1

36. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs), for Subjects in the Flu Vaccine Cohort
Description: An unsolicited AE = any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. AEs were collected for subjects receiving Nimenrix vaccine lot A+Fluarix vaccine, Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: From Dose 1 (at Month 0) up to 1 month after vaccination (at Month 1)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 311 | 104
Participants | 13 | 50 | 20

37. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs), for Subjects in the Flu Vaccine Cohort
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. SAEs were collected for subjects receiving Nimenrix vaccine lot A co-administered with Fluarix vaccine, on subjects receiving Nimenrix vaccine (pooled groups from the Flu vaccine cohort) and on subjects receiving Mencevax ACWY vaccine (in the Flu vaccine cohort).
Time Frame: From Dose 1 (at Month 0) up to study end (at Month 6)
Population: The Total Vaccinated Cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix (Flu Cohort) Group: Group Nimenrix A Group, Nimenrix B Group and Nimenrix C Group pooled groups from the Flu vaccine cohort. Nimenrix™ vaccine was administered by intramuscular injection in the deltoid region of the non-dominant arm.
Arm/Group | Nimenrix+Fluarix Group | Nimenrix (Flu Cohort) Group | Mencevax ACWY (Flu Cohort) Group
Number analyzed (Participants) | 105 | 311 | 104
Participants | 0 | 4 | 0

ADVERSE EVENTS:
Time Frame: SAEs: from Dose 1 at Month 0 up to study end at Month 6. Solicited local and general symptoms: During the 4-day (Days 0-3) post-vaccination period after vaccination.
Description: The number of subjects reporting solicited local symptoms in the Nimenrix+Fluarix Group was tabulated for any vaccination. Among the 105 subjects of the group, 23, 6 and 4 subjects reported pain, redness and swelling post-meningococcal vaccination and 29, 7 and 7 subjects reported pain, redness and swelling post-Fluarix vaccination.
Arm/Group | Nimenrix Group | Mencevax ACWY Group | Nimenrix+Fluarix Group
All-Cause Mortality (participants affected / at risk) | 0/935 | 0/312 | 0/105
Serious Adverse Events (participants affected / at risk) | 7/935 | 1/312 | 0/105
Other Adverse Events (participants affected / at risk) | 330/935 | 89/312 | 49/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix Group (N=935) | Mencevax ACWY Group (N=312) | Nimenrix+Fluarix Group (N=105)
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix Group (N=935) | Mencevax ACWY Group (N=312) | Nimenrix+Fluarix Group (N=105)
Pain (General disorders) | 180 | 42 | 37
Redness (General disorders) | 82 | 14 | 11
Swelling (General disorders) | 73 | 6 | 10
Fatigue (General disorders) | 114 | 30 | 10
Headache (General disorders) | 151 | 44 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.